CLINICAL TRIAL: NCT03171012
Title: Proprioceptive Neuromuscular Facilitation Repercussions Associated With Cardiorespiratory Training in Postal Individuals Stroke to the Functions Motor, Respiratory and Quality of Life: Randomized Controlled Trial
Brief Title: Addition of Proprioceptive Neuromuscular Facilitation to Cardio Respiratory Training Post Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Renata Janaína Pereira de Souza, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LACAP UFPE/UFRN
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Chest Wall Disorder; Quality of Life
Keywords: Muscle Stretching Exercises
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises; Respiration

STUDY DESIGN:
Intervention Model Description: Forty individuals into four groups: Experimental Lower Limbs (LL's CRT with PNF); Group control Lower Limbs (LL's CRT with respiration). Experimental Upper Limbs (UP's CRT with PNF) and Group control Upper Limbs (UP's CRT with respiration). Individuals will be assessed before and immediately after 20 program sessions and one month after the end of treatment.
  The treatment program will have the full duration of One hour including: ten minutes of stretching (five minutes before and five Minutes after the therapeutic intervention), ten minutes of rest and 40 minutes of Aerobic treatment associated with PNF or to respiration, being performed in 20 Sessions three times a week. For therapy with the CRT used the cycle ergometer for lower or upper limbs, Based on the criteria of the ACSM and monitoring Constant blood pressure, oxygen saturation and perceived exertion. The PNF patterns will be performed in seated, dorsal, ventral and Side.
Who Masked: Participant, Investigator
Masking Description: Randomization will be by randomization.com software, where a third person, who will not participate in the other stages of the survey, execute the process and deliver the opaque and numbered envelopes to the researcher responsible for the training, thus ensuring the confidentiality of the allocation. The patient may be allocated to the LL's CRT + PNF group, LL's CRT + Breathing, UL's CRT + PNF or UL's CRT + Breathing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lower limbs CRT+ PNF (Experimental): Lower Limbs Cardiorespiratory training associated with Proprioceptive Neuromuscular Facilitation
  Interventions: Other: Lower limbs CRT; Other: Proprioceptive Neuromuscular Facilitation
- Lower limbs CRT + respiration (Active Comparator): Lower limbs Cardiorespiratory training associated with respiration
  Interventions: Other: Lower limbs CRT; Other: respiration
- Upper limbs CRT + PNF (Experimental): Upper limbs Cardiorespiratory training associated with Proprioceptive Neuromuscular Facilitation
  Interventions: Other: Upper limbs CRT; Other: Proprioceptive Neuromuscular Facilitation
- Upper limbs CRT + respiration (Active Comparator): Upper limbs Cardiorespiratory training associated with respiration
  Interventions: Other: Upper limbs CRT; Other: respiration

INTERVENTIONS:
Other: Lower limbs CRT — cycle ergometer for lower limbs
  Arms: Lower limbs CRT + respiration; Lower limbs CRT+ PNF
Other: Upper limbs CRT — cycle ergometer for upper limbs
  Arms: Upper limbs CRT + PNF; Upper limbs CRT + respiration
Other: Proprioceptive Neuromuscular Facilitation — Proprioceptive Neuromuscular Facilitation patterns will be performed in seated, dorsal, ventral and side.
  Arms: Lower limbs CRT+ PNF; Upper limbs CRT + PNF
Other: respiration — respiration
  Arms: Lower limbs CRT + respiration; Upper limbs CRT + respiration

SUMMARY:
Post-stroke hemiparesis causes sequelae in the limbs and also in the trunk and abdomen structures. The level of physical activity decreases and cardiorespiratory training(CRT) is indicated to this population to improve the functions of several systems (respiratory, cardiovascular, muscular). The application of Proprioceptive Neuromuscular Facility(PNF) would imply in the awareness and greater harmony of the functions performed by the trunk of this individual. The objective of this study is to evaluate the effects of respiratory and trunk characteristics of the PNF associated with Cardiorespiratory training in quality of life, gait, distance traveled, peak oxygen consumption, respiratory muscle strength, thoracic cavity volumes, mobility and diaphragmatic thickness of individuals with post stroke.

DETAILED DESCRIPTION:
Clinical, randomized, blind and allocation. Forty individuals post-stroke will be randomized into four groups: Experimental Lower Limbs(submitted to LL's CRT associated with PNF); Group control Lower Limbs (submitted LL's CRT associated with respiration). Experimental Upper Limbs (submitted to UP's CRT associated with PNF) and Group control Upper Limbs (submitted to UP's CRT associated with respiration). Individuals will be assessed before and immediately after 20 program sessions and one month after the end of treatment. Outcome measures shall be measured by: Stroke Specific Quality of Life Scale; Inertial gear sensor; Maximum volume of oxygen; Spirometry and manovacuometry; Ultrasound of mobility and thickness diaphragmatic; compartmental volumes of the rib cage with opto plethysmography electronics.

For the four groups, the treatment program will have the total duration of one hour including: ten minutes of stretching (five minutes before and five minutes after the therapeutic intervention), ten minutes of rest and 40 minutes of aerobic treatment associated to PNF or to respiration, being performed in 20 Sessions three times a week. The order of application of the techniques will be random, being held until the end of the intervention period. For therapy with the CRT used the cycle ergometer for lower or upper limbs, Based on the criteria of the American College of Sports Medicine and monitoring constant blood pressure, oxygen saturation and perceived exertion. The PNF patterns will be performed in seated, dorsal, ventral and side. The breathing exercises will be performed at the same time and in the positions of the PNF. To analyze the data and to achieve the objectives appropriate statistical tests shall be used, according to the normality of and characteristics of the variables.

ELIGIBILITY:
Inclusion Criteria:

* Have clinical diagnosis of ischemic or hemorrhagic stroke,
* primary for more than six months resulting in hemiparesis;
* Have mental competence assessed through the Mini-Exam of the Mental State-MMSE;
* Be able to walk 10 meters independently, with or without assistive device;
* Absence of other neurological or orthopedic deficiencies unrelated to stroke;
* Without report of associated pulmonary pathology and not be smoker or ex-smoker.

Exclusion Criteria:

-

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen uptake | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  maximum oxygen volume consumed during the 6-minute walk test
Balance | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  The scale assesses the balance based on 14 common items of day-to-day.
Quality of life | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  12 domains: Energy (3 items); Family Relationships (3 items); Language (5 items); Mobility (6 items); Mood (5 items); Personality (3 items); Self-Care (5 items), Superior Member Function (5 items), Social Relations (5 items), Memory / Concentration (3 items), Vision (3 items) and Work / Productivity (3 items).
Gait | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Wireless system consisting of an inertial sensor, consisting of a 3-axis accelerometer, a magnetic sensor and a 3-axis gyroscope, which positioned in L5 allows a functional gait analysis. The system calculates from the data obtained all the temporal and spatial gait parameters required to perform a diagnosis or to define a training strategy. The distance traveled, time of support and balance, step size.
Compartmental volumes of the rib cage | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Analysis of the kinematics of the thoracic wall through the optical-electronic plethysmograph

SECONDARY OUTCOMES:
Respiratory function | Three months total:After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Spirometry: Will be measured slow vital capacity (Measured in liters), Inspiratory capacity (Measured in liters), forced expiratory volume in the first second (Measured in liters), Forced vital capacity (Measured in liters), forced expiratory volume ratio in the first second by forced vital capacity, peak expiratory flow (Measured in liters per minute).
Inspiratory muscle strength | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Manovacuometry: Maximal Inspiratory pressure (MIP), Measured in centimeters of water
Expiratory muscle strength | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Manovacuometry: maximal expiratory pressure (MEP), Measured in centimeters of water
Diaphragmatic thickness | Three months total: After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Measurement of the diaphragmatic thickness from the middle of the pleural line to the middle of the peritoneal line.
Mobility diaphragmatic | Three months total:After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  Using convex transducer (3.5MHz) positioned in the right axillary line below the costal margin, the examiner will maintain a firm hand towards the cranial direction. The cranio-caudal excursions of the diaphragm during quiet and forced breathing will record sinusoidal curves, which will represent the diaphragmatic mobility when the trajectory between the baseline at the beginning of the inspiration and the line obtained at the peak of the inspiration is verified.
Oxygen Uptake Efﬁciency Slope | Three months total:After 20 sessions of intervention(2 months) and after 1 months without treatment (follow-up)
  The OUES reﬂects the relationship between oxygen uptake(˙VO 2 in ml/min) and total ventilation (VE in L/min) and is best described by a single exponential function in almost all subjects.
  This index was determined by the following equation: VO2 = a log10VE + b When VO 2 in ml/min is plotted on the y axis and VE in L/min is plotted on the semilog transformed x axis, the slope of this linear relationship, "a", represents the OUES.

CONTACTS AND LOCATIONS:
Overall Officials: RENATA SOUZA, MASTER, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Souza RJP, Brandao DC, Martins JV, Fernandes J, Dornelas de Andrade A. Addition of proprioceptive neuromuscular facilitation to cardiorespiratory training in patients poststroke: study protocol for a randomized controlled trial. Trials. 2020 Feb 14;21(1):184. doi: 10.1186/s13063-019-3923-1. PMID 32059691